CLINICAL TRIAL: NCT04370509
Title: A Phase II Study of Perioperative Pembrolizumab-Based Therapy in Patients With Locally Advanced or Metastatic Renal Cell Carcinoma Prior to Cytoreductive Nephrectomy or Metastasectomy
Brief Title: Pembrolizumab With or Without Axitinib for Clear Cell Kidney Cancer in Patients Undergoing Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Collaborating sponsor decision
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 197017; NCI-2020-02128 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma; Recurrent Clear Cell Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell | interventions — Axitinib; Cytoreduction Surgical Procedures; Nephrectomy; Metastasectomy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Pembrolizumab monotherapy) (Experimental): Preoperative treatment consists of 200mg pembrolizumab IV on day 1 of each cycle. Treatment repeats every 21 days for up to 3 cycles (9 weeks).
  Within 14-21 days following the end of treatment, patients undergo standard of care CN or MET. Patients with PD may undergo CN or MET per physician discretion.
  Within 21-42 days after surgery, patients with R0 resection or R1 resection receive 400 mg pembrolizumab every 42 days for up to 9 cycles (1 year) and patients with R2 resection receive pembrolizumab every 42 days for up to 18 cycles (2 years) in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Cytoreductive Nephrectomy (CN); Procedure: Metastasectomy (MET); Biological: Pembrolizumab
- Cohort B (Pembrolizumab + VEGF-TKI) (Experimental): Preoperative treatment consists of 200 mg pembrolizumab IV on day 1 of each cycle, and 5mg axitinib (a vascular endothelial growth factor (VEGF) tyrosine kinase inhibitor (TKI)) PO BID on days 1-42 of each cycle. Axitinib maybe titered in select patients after cycle 1. Treatment repeats every 21 days for up to 3 cycles (9 weeks).
  Within 14-21 days following the end of pre-operative treatment, patients undergo standard of care CN or MET. Patients with PD may undergo CN or MET per physician discretion.
  Within 21-42 days after surgery, patients with an R0 or R1 resection receive 400 mg pembrolizumab and 1, 3, 5, 7 or 10 mg axitinib PO BID every 42 days for up to 9 cycles (1 year), and patients with an R2 resection receive pembrolizumab IV and axitinib PO BID every 42 days for up to 18 cycles (2 years) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Axitinib (VEGF-TKI); Procedure: Cytoreductive Nephrectomy (CN); Procedure: Metastasectomy (MET); Biological: Pembrolizumab

INTERVENTIONS:
Drug: Axitinib (VEGF-TKI) — Given PO
  Other Names: AG-013736; AG013736; Inlyta
  Arms: Cohort B (Pembrolizumab + VEGF-TKI)
Procedure: Cytoreductive Nephrectomy (CN) — Undergo CN
  Other Names: Cytoreduction; Nephrectomy
Procedure: Metastasectomy (MET) — Undergo MET
  Other Names: Metastasectomy
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab with or without standard of care axitinib works in treating patients with clear cell kidney cancer that has spread to nearby tissues or lymph nodes (locally advanced) or other places in the body (metastatic) who are undergoing surgery. Pembrolizumab is an antibody that is designed to bind to and block the activity of PD-1, a molecule in the body that may be responsible for inhibiting the body's immune response against cancer cells. Axitinib is a type of drug known as a tyrosine kinase inhibitor. Tyrosine kinase inhibitors work by blocking enzymes called tyrosine kinases. These enzymes may be too active or found at high levels in some types of cancer cells and blocking them may help keep cancer cells from growing. Giving pembrolizumab with or without axitinib may work better in controlling the cancer and decrease the likelihood of it coming back following surgery in patients with kidney cancer compared to usual treatment (surgery followed by chemotherapy and/or radiation therapy).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the impact of pembrolizumab-based therapy on the composition, phenotype, and function of tumor-infiltrating immune cells (TIICs) in subjects with advanced renal cell carcinoma (RCC) undergoing cytoreductive nephrectomy (CN)/metastasectomy (MET).

SECONDARY OBJECTIVES:

I. To determine the clinical efficacy of preoperative pembrolizumab-based therapy in subjects with advanced RCC undergoing CN/MET.

II. To explore the clinical efficacy of continued pembrolizumab-based therapy following CN/MET in subjects with advanced RCC.

III. To determine the safety and tolerability of pembrolizumab-based therapy in subjects with advanced RCC undergoing CN/MET.

EXPLORATORY OBJECTIVES:

I. To explore the clinical efficacy of preoperative pembrolizumab-based therapy in subjects with advanced RCC, by pathologic response. (Clinical).

II. To explore the relationship between changes in TIICs and clinical efficacy in subjects with advanced RCC treated with pembrolizumab-based therapy. (Scientific).

III. To characterize changes in the frequency and number of circulating T cells induced by pembrolizumab-based therapy in subjects with advanced RCC. (Scientific).

IV. To determine the impact of pembrolizumab-based therapy on the composition and phenotype of the tumor microenvironment (including tumor and stromal cells) in subjects with advanced RCC. (Scientific).

V. To determine whether locally advanced versus metastatic RCC exhibit differences in immune composition or phenotype at baseline and in response to pembrolizumab-based therapy. (Scientific).

VI. To determine the change in T cell repertoire within the tumor and blood induced by pembrolizumab-based therapy in subjects with advanced RCC. (Scientific).

VII. To explore molecular profiles to identify potentially predictive biomarkers for subjects with advanced RCC treated with immunotherapy (Scientific).

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Within 14-21 days following the end of treatment, patients will undergo standard of care CN or MET. Patients with progressive disease (PD) may undergo CN or MET per physician discretion. Within 21-42 days after surgery, patients with no disease (R0 resection) or microscopic disease (R1 resection) receive pembrolizumab IV every 42 days for up to 9 cycles (1 year) and patients with macroscopic disease (R2 resection) receive pembrolizumab IV every 42 days for up to 18 cycles (2 years) in the absence of disease progression or unacceptable toxicity

COHORT B: Patients receive pembrolizumab IV over 30 minutes on day 1 and standard of care axitinib orally (PO) twice daily (BID) on days 1-42. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Within 14-21 days following the end of treatment, patients undergo standard of care CN or MET. Patients with PD may undergo CN or MET per physician discretion. Within 21-42 days after surgery, patients with an R0 or R1 resection receive pembrolizumab IV over 30 minutes on day 1 and axitinib PO BID on days 1-42. Treatments repeat every 42 days for up to 9 cycles (1 year) in the absence of disease progression or unacceptable toxicity. Patients with an R2 resection receive pembrolizumab IV over 30 minutes on day 1 and axitinib PO BID on days 1-42. Treatment repeats every 42 days for up to 18 cycles (2 years) in the absence of disease progression or unacceptable toxicity.

Follow-up will occur at treatment discontinuation, 30 days post-discontinuation, and then every 12 weeks for up to 1 year post-discontinuation. Subjects who discontinue study participation due to progressive disease will return for a mandatory safety follow-up visit within 30 days of(+7 days) after the final dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed RCC with a clear cell component.
2. Locally advanced or metastatic disease (primary intact or status post nephrectomy with recurrent disease)
3. Planned CN and/or MET.
4. Must have a tumor lesion amenable to biopsy at pre-treatment and subjects must consent to acquisition of fresh tumor specimens obtained using the following approaches:

   1. Core biopsy.
   2. Nephrectomy.
   3. Metastasectomy (MET). Note: Subjects who undergo nephrectomy or metastasectomy prior to study enrollment must still have measurable disease (RECIST 1.1) that is amenable to cytoreductive nephrectomy or metastasectomy to be eligible for study participation.
   4. Fine needle aspiration (FNA) specimens are not acceptable.
5. Measurable disease per RECIST 1.1 as assessed by the investigator. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Subject (or legally acceptable representative if applicable) must provide written informed consent for the trial.
7. At least 18 years of age on day of signing informed consent.
8. Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
9. Adequate organ function as defined in Table 1; all screening labs should be performed within 10 days of treatment initiation.

   1. Absolute neutrophil count (ANC) >= 1,500/microliter (uL)
   2. Platelets >= 100,000/uL.
   3. Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment).
   4. Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (CrCl) (glomerular filtration rate (GFR) can also be used in place of creatinine or CrCl) >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN. Creatinine clearance should be calculated per institutional standard.
   5. Serum total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 ULN.
   6. Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT)) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 2.5 x ULN.
   7. Albumin >= 2.5 mg/dL.
   8. International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants.
   9. Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (within 10 days of treatment initiation)
10. Negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication (day 1) (female participants of childbearing potential). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
11. Male and female participants of childbearing potential must be willing to use an adequate method of contraception* for the course of the study through 120 days after the last dose of study medication. * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

1. RCC WITHOUT a clear cell component.
2. Prior systemic therapy for the treatment of RCC.
3. No measurable disease (e.g. only bone metastases).
4. Not a candidate for CN and/or MET.
5. Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks since the last dose of the previous investigational agent
6. Diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
7. Known history of active Bacillus tuberculosis (TB).
8. Severe hypersensitivity (>= grade 3) to pembrolizumab/axitinib or any of their excipients.
9. Prior systemic anti-cancer monoclonal antibody (mAb), targeted small molecule therapy, or radiation therapy within 2 weeks prior to the first dose of study treatment (Day 1).

   * Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline. Participants with =< grade 2 neuropathy may be eligible.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
   * Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
10. Known additional malignancy that is progressing or has required active treatment within the past 2 years.

    * Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
11. Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
12. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
13. History of (non-infectious) pneumonitis that required treatment with steroids or has current pneumonitis.
14. Active infection requiring systemic therapy.
15. Any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to randomization.
16. Uncontrolled or poorly controlled hypertension despite standard medical therapy.
17. Serious or nonhealing wound, ulcer, or bone fracture within 28 days of study enrollment.
18. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
19. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
20. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
21. Any prior therapy with an anti-PD-1, anti-PD-L1,or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137).
22. Known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
23. Known history of hepatitis B (defined as hepatitis B surface antigen reactive) or known active hepatitis C virus (defined as hepatitis C virus (HCV) ribonucleic acid (RNA) [qualitative] is detected) infection. No testing for hepatitis B and hepatitis C is required unless mandated by local health authority.
24. Live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed.
25. History of grade 3-4 gastrointestinal (GI) bleeding within 12 weeks prior to study enrollment.
26. Solid organ or hematologic transplant.
27. Encephalopathy in the last 6 months. Those participants on rifaximin or lactulose to control their encephalopathy are not allowed.
28. Evident ascites on physical examination.

    * Note: Medically controlled ascites and ascites detectable on imaging studies only is allowed
29. Female of childbearing potential who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
30. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Y Oh, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was closed to enrollment by the sponsor before enrollment in Cohort B was made available to participants. Therefore, no participants could be enrolled in Cohort B.
Groups:
- Cohort A (Pembrolizumab Monotherapy): Preoperative treatment consists of 200mg pembrolizumab IV on day 1 of each cycle. Treatment repeats every 21 days for up to 3 cycles (9 weeks).
  Within 14-21 days following the end of treatment, patients undergo standard of care CN or MET. Patients with progressive disease (PD) may undergo CN or MET per physician discretion.
  Within 21-42 days after surgery, patients with R0 resection or R1 resection receive 400 mg pembrolizumab every 42 days for up to 9 cycles (1 year) and patients with R2 resection receive pembrolizumab every 42 days for up to 18 cycles (2 years) in the absence of disease progression or unacceptable toxicity.
- Cohort B (Pembrolizumab + VEGF-TKI): Preoperative treatment consists of 200 mg pembrolizumab IV on day 1 of each cycle, and 5mg axitinib (a vascular endothelial growth factor (VEGF) tyrosine kinase inhibitor (TKI)) orally (PO) twice a day (BID) on days 1-42 of each cycle. Axitinib maybe titered in select patients after cycle 1. Treatment repeats every 21 days for up to 3 cycles (9 weeks).
  Within 14-21 days following the end of pre-operative treatment, patients undergo standard of care CN or MET. Patients with PD may undergo CN or MET per physician discretion.
  Within 21-42 days after surgery, patients with an R0 or R1 resection receive 400 mg pembrolizumab and 1, 3, 5, 7 or 10 mg axitinib PO BID every 42 days for up to 9 cycles (1 year), and patients with an R2 resection receive pembrolizumab IV and axitinib PO BID every 42 days for up to 18 cycles (2 years) in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort A (Pembrolizumab Monotherapy) | Cohort B (Pembrolizumab + VEGF-TKI)
Started | 6 | 0
Completed Cytoreductive Nephrectomy (CN) or Metastasectomy (MET) | 5 | 0
Received 1 Year of Pembrolizumab | 4 | 0
Completed | 4 | 0
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Did not receive post-op Pembrolizumab | 1 | 0

BASELINE CHARACTERISTICS:
Population: The study was closed by the sponsor to further enrollment before Cohort B was open for accrual.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Pembrolizumab Monotherapy) | Cohort B (Pembrolizumab + VEGF-TKI) | Total
Number analyzed (Participants) | 6 | 0 | 6
Age, Customized [Count of Participants; unit: Participants]
  40-49 years old | 1 | 0 | 1
  50-59 years old | 1 | 0 | 1
  60-69 years old | 1 | 0 | 1
  70-79 years old | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 2 | 0 | 2
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 0 | 3
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 |  | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With >= 2-fold Increase in the Number of Tumor-infiltrating Immune Cells (TIICs)
Description: TIICs will be analyzed in pre- and post-pembrolizumab-based treatment tumor specimens. The proportion of participants with a >=2-fold increase (from pre- to post-treatment) in the number of TIICs will be calculated.
Time Frame: Baseline to cytoreductive nephrectomy (CN)/metastasectomy (MET), up to 1 year
Population: The analysis for this endpoint could not be completed due to insufficient funds for the laboratory experiments to determine the number of tumor-infiltrating immune cells (TIICs), when the collaborating sponsor (Merck Sharp and Dohme) terminated the study prematurely. Therefore, no plans currently exist to fund analysis of this endpoint in the future.
Arm/Group | Cohort A (Pembrolizumab Monotherapy)
Number analyzed (Participants) | 0

2. Secondary Outcome: Objective Response Rate (ORR) in Pre-operative Pembrolizumab-based Therapy
Description: Objective response rate in pre-operative pembrolizumab-based therapy in participants with advanced renal cell carcinoma (RCC) will be defined as proportion of participants who obtain a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors 1.1 modified to allow a maximum of 10 target lesions or 5 target lesions per organ. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm; Partial Response (PR), >=At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; Overall Response (OR) = CR + PR.
Time Frame: Up to 1 year
Measure: Number; unit: proportion of participants
Arm/Group | Cohort A (Pembrolizumab Monotherapy)
Number analyzed (Participants) | 6
proportion of participants | 0

3. Secondary Outcome: Disease-Free Survival Rate (DFS) at 1 Year for Participants Who Obtain CR or PR/SD With R0 Resection and Are Treated 1 Year of Pembrolizumab-based Therapy
Description: The DFS for continued pembrolizumab-based therapy in participants with advanced RCC will be assessed in participants who achieve CR, PR, or stable disease (SD) followed by R0 resection, and is defined as the proportion of those participants who remain disease-free at the end of the 1 year continued treatment period (1-year DFS rate)
Time Frame: Up to 1 year
Measure: Number; unit: proportion of participants
Arm/Group | Cohort A (Pembrolizumab Monotherapy)
Number analyzed (Participants) | 4
proportion of participants | 1.0

4. Secondary Outcome: Disease-Free Survival Rate (DFS) at 2 Years for Participants Who Obtain CR or PR/SD With R0 Resection and Are Treated 1 Year of Pembrolizumab-based Therapy
Description: The DFS for continued pembrolizumab-based therapy in participants with advanced RCC will be assessed in participants who achieve CR, PR, or stable disease (SD) followed by R0 resection, and is defined as the proportion of those participants who remain disease-free at 1 year following the end of the continued treatment period (2-year DFS rate)
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Cohort A (Pembrolizumab Monotherapy)
Number analyzed (Participants) | 4
proportion of participants | 0.5

5. Secondary Outcome: Median DFS for Participants Who Obtain CR or PR/SD With R0 Resection and Are Treated 1 Year of Pembrolizumab-based Therapy
Description: In participants who achieve CR, PR or stable disease (SD) followed by R0 resection, median time participants remain disease-free will be reported using the Kaplan-Meier estimate.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort A (Pembrolizumab Monotherapy)
Number analyzed (Participants) | 4
days | 651 [602 to NA] — There were insufficient number of events so the upper limit could not be reached.

6. Secondary Outcome: Progression-free Survival Rate (PFS) at 1 Year for Participants Who Obtain PR/SD and Have Residual Disease Following CN/MET and Are Treated With 1 Year of Pembrolizumab-based Therapy
Description: PFS for participants who achieve PR/SD with residual disease following CN/MET and are also treated with 1 year of pembrolizumab-based therapy is defined as the proportion of participants who remain progression-free at the end of the 1 year continued treatment period (1-year PFS rate)
Time Frame: Up to 1 year
Population: No participants achieved PR/SD with residual disease; therefore, data were not collected from any participants.
Arm/Group | Cohort A (Pembrolizumab Monotherapy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Progression-free Survival Rate (PFS) at 2 Years for Participants Who Obtain PR/SD and Have Residual Disease Following CN/MET and Are Treated With 1 Year of Pembrolizumab-based Therapy
Description: PFS in participants who achieve PR/SD with residual disease following CN/MET and are also treated with 1 year of pembrolizumab-based therapy is defined as the proportion of participants who remain progression-free at 1 year following the end of the continued treatment period (2-year PFS rate)
Time Frame: Up to 2 years
Population: No participants achieved PR/SD with residual disease; therefore, data were not collected from any participants.
Arm/Group | Cohort A (Pembrolizumab Monotherapy)
Number analyzed (Participants) | 0

8. Secondary Outcome: Median PFS for Participants Who Obtain PR/SD and Have Residual Disease Following CN/MET and Are Treated With 1 Year of Pembrolizumab-based Therapy
Description: The Median PFS for participants who obtain PR/SD and have residual disease following CN/MET and are treated with 1 year of pembrolizumab-based therapy will be reported as the median time participants remain progression-free using the Kaplan-Meier estimate.
Time Frame: Up to 2 years
Population: No participants achieved PR/SD with residual disease; therefore, data were not collected from any participants.
Arm/Group | Cohort A (Pembrolizumab Monotherapy)
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants Reporting Treatment-related Adverse Events
Description: Adverse events classified as being definitely, possibly, or probably related to study treatment will be assessed and reported using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Pembrolizumab Monotherapy)
Number analyzed (Participants) | 6
Participants | 6

10. Secondary Outcome: Number of Participants Reporting Surgical Complications
Description: The number of participants reporting surgical complications by grade using the Clavien-Dindo Classification of Surgical Complications will be reported.
Time Frame: Up to 2 years
Population: One participant withdrew from the study prior to receiving surgery and was excluded from this endpoint analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Pembrolizumab Monotherapy)
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Cohort A (Pembrolizumab Monotherapy)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Pembrolizumab Monotherapy) (N=6)
Colitis (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Pembrolizumab Monotherapy) (N=6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (7)
Fatigue (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Creatinine increased (Investigations) | 3 (4)
Weight loss (Investigations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (4)
Hematuria (Renal and urinary disorders) | 2 (3)
Myocarditis (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated earlier than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT04370509/Prot_SAP_000.pdf